CLINICAL TRIAL: NCT06996522
Title: Underwater Endoscopic Mucosal Resection Versus Hot Snare Polypectomy in the Treatment of Pedunculated Colorectal Polyps Less Than 10mm in Size: A Single-center, Open-label, Randomized Controlled Trial
Brief Title: UEMR Versus HSP in the Treatment of Pedunculated Colorectal Polyps Less Than 10mm in Size
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025K132
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pedunculated Colorectal Polyp
Keywords: Pedunculated colorectal polyp; Underwater endoscopic mucosal resection; Hot snare polypectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UEMR in treating Pedunculated colorectal polyps less than 10mm in size (Experimental): The UEMR procedure included the following: (1) Water infusion to distend the intestinal lumen; (2) entrapment of the mucosal protrusion with a snare; and (3) resection using electrocautery
  Interventions: Procedure: underwater endoscopic mucosal resection
- HSP in treating Pedunculated colorectal polyps less than 10mm in size (Active Comparator): The HSP procedure included the following: (1) entrapment and resection of the polyp with a snare with electrocautery.
  Interventions: Procedure: Hot snare polypectomy

INTERVENTIONS:
Procedure: underwater endoscopic mucosal resection — The Pedunculated colorectal polyps less than 10mm in size in this group will be treated by UEMR
  Arms: UEMR in treating Pedunculated colorectal polyps less than 10mm in size
Procedure: Hot snare polypectomy — The Pedunculated colorectal polyps less than 10mm in size in this group will be treated by HSP
  Arms: HSP in treating Pedunculated colorectal polyps less than 10mm in size

SUMMARY:
A prospective, single-center, open-label, randomized controlled study to compare the effectiveness and safety of underwater endoscopic mucosal resection (UEMR) and hot snare polypectomy (HSP) in treating Pedunculated colorectal polyps less than 10mm in size.

DETAILED DESCRIPTION:
1. Patients are undergone screening, surveillance, or therapeutic colonoscopy at the Endoscopy department of Gastrointestinal endoscopy center of Huadong hospital affiliated to Fudan University.
2. Randomize patients with pedunculated colorectal polyps less than 10mm in size into 2 interventional groups based on Random function of Statistical Package for the Social Sciences (SPSS) 20.0, including (1) Group 1: Underwater endoscopic mucosal resection (UEMR) and (2) Group 2: Hot snare polypectomy (HSP).
3. Collecting variables which consist of primary and secodary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 35 and 80 years
* Pedunculated colorectal polyps less than 10mm in size in screening, surveillance or therapeutic colonoscopy
* 0-Isp or 0-Ip according to Paris classification
* Patients must sign an informed consent form prior to registration in study

Exclusion Criteria:

* Unsuitable for removal by UEMR or HSP
* Suspected malignancy
* History of inflammatory bowel disease or colorectal resection
* Familial adenomatous polyposis or Lynch syndrome
* Patients taking anticoagulant and antiplatelet agents before the examination
* Inadequate bowel preparation, defined as a Boston Bowel Preparation Scale score < 6
* ASA >=3
* Pregnancy or breastfeeding
* Severe comorbid disease involving the heart, lungs, liver, or kidneys.
* Concurrent serious conditions, including other active malignancies or severe infectious diseases

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Post-polypectomy Bleeding | 2 weeks after the procedure
  Presence of Clinically Significant Immediate Post-polypectomy Bleeding（CSIPB） or Clinically Significant Delayed Post-polypectomy Bleeding (CSDPB). CSIPB was defined as any bleeding not responding to water jet irrigation or STSC and therefore requiring either coagu lation forceps or mechanical clips to achieve hemostasis. CSDPB was defined as any bleeding after completion of the procedure requiring emergency room presentation, hospital isation or re-intervention (endoscopy, angiography, surgery).

SECONDARY OUTCOMES:
postoperative electrocoagulation syndrome | 2 weeks after the procedure
  Postoperative electrocoagulation syndrome （PEECS）defined as localized abdominal tenderness plus at least one of the following: (1) body temperature > 37.6 °C; (2) white-blood-cell count > 10 × 10⁹ /L; or (3) C-reactive protein > 0.5 mg/dL, after ruling out delayed postoperative perforation).
en bloc resection | immediately after the procedure
  Rate of en bloc resection rate
R0 resection | 2 weeks after the procedure
  Rate of R0 resection
Delayed perforation | 2 weeks after the procedure
  Rate of delayed perforation

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyu Dong, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital affiliated to Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: 18817870866@163.com)